CLINICAL TRIAL: NCT02422329
Title: Changes in Patient Reported Constipation Among Advanced Cancer Patients After Receiving an Educational Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0111; NCI-2015-00734 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Constipation; Recurrent cancer; Locally advanced cancer; Metastatic cancer; Video; Fact sheet; Questionnaires; Surveys
MeSH Terms: conditions — Constipation; Recurrence; Neoplasm Metastasis | interventions — Surveys and Questionnaires; Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Video (Experimental): Participants complete self-administered numerical rating scale (NRS) constipation questionnaire at baseline. Participants watch a 3-minute educational video describing symptoms of constipation and importance of regular bowel movements. Participants then complete three self-administered questionnaires, post-educational material, Modified Rome III questionnaire, and Overall satisfaction of the educational material.
  Interventions: Behavioral: Questionnaires; Behavioral: Video
- Fact Sheet (Experimental): Participants complete self-administered numerical rating scale (NRS) constipation questionnaire at baseline. Participants read educational material describing symptoms of constipation and importance of regular bowel movements. Participants then complete three self-administered questionnaires, post-educational material, Modified Rome III questionnaire, and Overall satisfaction of the educational material.
  Interventions: Behavioral: Questionnaires; Behavioral: Fact Sheet

INTERVENTIONS:
Behavioral: Questionnaires — Participants complete questionnaires at baseline and after intervention.
  Other Names: Surveys
Behavioral: Video — Participants watch a 3-minute educational video describing symptoms of constipation and importance of regular bowel movements.
  Arms: Educational Video
Behavioral: Fact Sheet — Participants read educational material describing symptoms of constipation and importance of regular bowel movements.
  Arms: Fact Sheet

SUMMARY:
The goal of this research study is to learn how patients' think about constipation before and after receiving education about the subject.

DETAILED DESCRIPTION:
If participant agrees to take part in the study, information about them (such as their age, gender, ethnicity, religion, diagnosis, and drugs they are currently taking) will be collected from their medical record.

Participant will also complete 1 questionnaire about constipation. It should take about 1-3 minutes to complete the questionnaire.

After completing the questionnaire, participant will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group. Participant will have an equal chance of being in either group.

* If participant is assigned to Group 1, they will watch a short educational video.
* If participant is assigned to Group 2, they will read a fact sheet.

Both the video and the fact sheet describe symptoms of constipation and the importance of regular bowel movements. They should take about 3 minutes each to complete.

After participant has viewed the educational material, they will complete 3 questionnaires about constipation and how helpful they think the video or fact sheet was in educating them about constipation. It should take about 10 minutes total to complete these questionnaires. Participant will watch the video/read the fact sheet and complete the questionnaires in their room at the Supportive Care Clinic.

Length of Study:

Patient's participation on this study will be over after they have completed the last 3 questionnaires.

This is an investigational study.

Up to 200 participants will be enrolled in the study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of advanced cancer, including recurrent, locally advanced, or metastatic cancer
2. Age >/= 18 years old
3. Patients must be able to understand, read, write, and speak English
4. Patients must have no clinical evidence of cognitive impairment as determined by the palliative care physician (Memorial Delirium Assessment Score >/= 7)
5. Patients must sign an informed consent

Exclusion Criteria:

1. Patients with a diagnosis of inflammatory bowel disease, i.e. Crohn's disease or ulcerative colitis
2. Patients with complete or partial bowel obstruction as determined by the palliative care physician
3. Patients with a bowel ostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Perception of Constipation | 1 day
  Primary objective is to examine effect of educational intervention on the patient-reported perception of constipation (PRC, by a 0-10 numeric rating score) among advanced cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org